CLINICAL TRIAL: NCT02862626
Title: Assessment of Psychological State of Mothers of Diabetic Children Aged 5 and Under (in Terms of Depression, Stress, Coping , Anxiety, Fear of Hypoglycemia) and Influencing Factors of This Psychological State
Acronym: PSY-DIA-MUM
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: P/2015/282
Record Dates: First submitted 2016-08-08; First posted 2016-08-11 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Depression
Keywords: Diabetic children; Mothers
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The incidence of type one diabetes is still rising, especially in children under 5 years old. Mothers often are the primary caregivers of these children. To take care of a young child with diabetes is a great responsibility and mothers must be constantly vigilant. This study aims to assess the psychological state of these mothers (in term of depression, anxiety, stress, coping, fear of hypoglycemia) and factors which influence this state.

ELIGIBILITY:
Inclusion Criteria:

* Mother of diabetic child aged 5 and under, followed-up in Pediatrics Department of Besançon University Hospital.

Exclusion Criteria:

* Mother of diabetic child older than 5 years old

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Mothers of diabetic children aged 5 and under followed-up in Pediatrics Department of Besançon University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2016-01-11 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of depression among mothers of children aged 5 or under with type 1 diabetes | at enrollment
  Assessment with self-administered questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte Mignot, MD, Principal Investigator — CHU Besançon
Locations (1):
- CHU Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: No